CLINICAL TRIAL: NCT05754554
Title: Clinical Study of Atlanto-occipital Decompression Lateral Joint Release Combined With Occipital-neck Fusion in the Treatment of Chiari Malformation Combined With Type II Skull Base Depression
Brief Title: Clinical Study of the Treatment of Chiari Malformation Combined With Type II Skull Base Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Yuntao Lu, Clinical Professor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2022-440
Record Dates: First submitted 2023-01-28; First posted 2023-03-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Atlantoaxial Dislocation; Chiari Malformation; Basilar Invagination
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Atlas occipital decompression lateral joint release combined with occipital-neck fusion — A. Chiari malformation combined with type II Basilar invagination showed that the slope spinal canal angle decreased, and the position of the dentition moved up. The yellow fusion device in the picture is C1/2 lateral inter-articular Cage (the patent granted by the applicant for this project); B. After atlanto-occipital decompression, C1/2 lateral inter-articular release is performed, and a fusion device is implanted to move down the position of the tip of the tooth process to reduce the compression of the cervical medulla oblongata; C. Implantation of the posterior neck nail rod system; D. Improve the angle of the sloped spinal canal by posterior compression rod technique (Cantilever) to further reduce the compression on the superior cervical medulla oblongata.

SUMMARY:
The research background of this study is that Chiari malformation (CM) is a congenital malformation in the foramen magnum region, often associated with syringomyelia, basilar depression, odontoid dislocation and other craniocervical junction deformities. The traditional surgical method for Chiari malformation with skull basilar depression is simple decompression without fixation, so it cannot effectively maintain the stability of the cervical spine and reduce the compression of the brainstem and cervical cord, often resulting in poor curative effect and aggravated symptoms. The cervical spine is the most flexible and most mobile part of the spine, and the instability of the cervical spine will directly affect the quality of life of patients after surgery. Subsequently, with the continuous advancement of technology and the continuous development and improvement of surgical methods, Investigators can relieve spinal cord compression by using atlanto-occipital decompression and dissection followed by C1/2 lateral arthrolysis combined with occipitocervical fusion. So, is this surgical combination the most effective surgery for patients with Chiari malformation and type II skull basilar depression? How should doctors adjust to the best surgical approach to treat patients with Chiari malformation and type II skull basilar depression? These questions have long puzzled neurosurgeons. By conducting this research, investigators hope that participants can participate in it, and work with them to answer this question, and jointly promote the development and progress of doctors' careers, while benefiting more patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chiari malformation
* Combined with type II skull base depression
* Clinical symptoms related to the disease
* Complete clinical imaging data
* Must be the first surgery

Exclusion Criteria:

* Secondary cerebellar tonsillar hernia
* Severe atlantoaxial dislocation
* Osteochondroplastica
* Rheumatoid arthritis
* Down syndrome
* Refurbished case reoperation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Chang of Chicago Chiari outcome score | through study completion, an average of 1 year
  The Chicago Chiari Malformation Prognosis Scale (CCOS) is a comprehensive quantitative scoring criterion for surgical prognosis in patients with Chiari malformations, first proposed by the Department of Neurosurgery of the University of Chicago School of Medicine. CCOS covered four scoring criteria, including improvement in pain symptoms, improvement in non-pain symptoms, ability to live, and surgery-related complications, with a single score of 1-4 for a total score of 4 to 16, and at the last follow-up, the higher the patient's score indicated the better the patient's postoperative prognosis.

SECONDARY OUTCOMES:
Occurrence of complications | The second week after surgery
  1)Minor complications such as pain, neck stiffness, and poor wound healing. 2)Serious complications such as vertebral artery injury, dyspnea, cerebrospinal fluid leakage, and severe intracranial infection.
Chang of Magnetic Resonance Imaging | through study completion, an average of 1 year
  Measurements of radiographic improvement, such as cerebellar tonsillar hernia length.
Chang of Visual Analog Score for pain | through study completion, an average of 1 year
  Visual Analog Score stands for visual analogue scoring method and is one of the commonly used pain scoring criteria. The main thing is to draw a 10cm horizontal line on the paper, the beginning end is 0, the other end is 10, the middle part represents different degrees of pain, let the patient choose the degree of pain by himself. A score below 3 represents mild pain; 4-6 are divided into pain that interferes with sleep, but is tolerable; A score of 7-10 indicates unbearable pain.
Chang of Japanese Orthopaedic Association Scores | through study completion, an average of 1 year
  The patient's lumbar spine function and improvement were mainly evaluated from four aspects: subjective symptoms, daily activity ability, clinical signs, and bladder function. The scoring range is 0~29 points, and the higher the total score, the milder the patient's condition.
Chang of Neck Disability Index | through study completion, an average of 1 year
  Neck Disability Index consists of 10 items, including: neck pain and related symptoms (pain intensity, headache, concentration and sleep) and activities of daily living (personal care, lifting heavy objects, reading, work, driving and playing). Each item has a minimum score of 0 and a maximum score of 5, with higher scores indicating greater levels of dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: yutao lu, Study Chair — 2Nanfang Neurology Research Institution, Nanfang Hospital, Southern Medical University
Locations (1):
- Nan fang hospital, Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No